CLINICAL TRIAL: NCT05005845
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Phase 2 Dose-Response Study to Determine Safety and Effectiveness of Two Concentrations of NFX-179 Gel in Subjects With Cutaneous Neurofibromas
Brief Title: NFX-179 Topical Gel Treatment for Adults With Neurofibromatosis 1 (NF1) and Cutaneous Neurofibromas (cNF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NFlection Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFX-179-NF1-202
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cutaneous Neurofibroma; Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5% NFX-179 gel (Active Comparator): Topical gel applied once daily to target cNFs
  Interventions: Drug: NFX-179 gel
- 1.5% NFX-179 gel (Active Comparator): Topical gel applied once daily to target cNFs
  Interventions: Drug: NFX-179 gel
- Vehicle gel (Placebo Comparator): Topical gel applied once daily to target cNFs
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: NFX-179 gel — NFX-179 topical gel is the active investigational product being studied
  Other Names: NFX-179 topical gel
  Arms: 0.5% NFX-179 gel; 1.5% NFX-179 gel
Drug: Vehicle gel — NFX-179 vehicle gel is the placebo comparator for this study
  Other Names: NFX-179 vehicle gel
  Arms: Vehicle gel

SUMMARY:
This is a randomized, double-blind, vehicle-controlled, parallel group dose response study evaluating the safety and effectiveness of 2 concentrations of NFX-179 Gel in subjects with cutaneous neurofibromas. At Visit 1, the investigator will identify 10 Target cNFs that fulfil the enrollment criteria. The Target cNFs must be located on the subject's face, anterior trunk, or upper extremities. Two Target cNFs must be on the face and 8 must be on the anterior trunk or upper extremities. The study medication will be applied topically QD to the Target cNFs for 182days (26 weeks). During the duration of the study subjects will be evaluated for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject must provide written informed consent prior to any study procedures
3. Subject must have a clinical diagnosis of NF1
4. Subject has 10 clinically diagnosed Target cNFs with preferably 2 Target cNFs located on the face and 8 Target cNFs located on the anterior trunk or upper extremities. Alternatively, at least 1 Target cNF is located on the face, in which case 9 Target cNFs must be located on the anterior trunk or upper extremities. Each Target cNF must meet the following criteria:

   * Has, in the investigator's opinion, a clinically typical appearance
   * Is not within 1 cm of the orbital rim
   * Is not covered with hair that might, in the investigator's opinion, interfere with obtaining photographs or impair evaluation of the cNF
   * Has a Physician's Tumor Assessment grade ≥2
   * Is dome shaped
   * Is not pedunculated
   * Is a discrete cNF surrounded by sufficient non-affected skin that, in the investigator's opinion:
   * The dimensions can be measured
   * The perimeter can be outlined in the study photographs
   * Is not irritated (e.g., bleeding, inflamed)
   * Is not in an area subject to repeated trauma (e.g., area that is shaved, on the beltline, under a bra strap, etc.)
   * Does not have an active cutaneous infection
   * Target cNFs on the face must have the following tumor dimensions:
   * Has a length that is ≥5mm and ≤14mm
   * Has a width that is ≥5mm and ≤14mm
   * Has a height that is ≥2mm.
   * Target cNFs on the anterior trunk or upper extremities must have the following tumor dimensions:
   * Has a length that is ≥7mm and ≤14mm
   * Has a width that is ≥5mm and ≤14mm
   * Has a height that is ≥2mm.
5. Subject agrees to avoid exposure of Target cNFs to excessive sunlight and to use her/his routine sunscreen if excessive exposure cannot be avoided
6. Subject agrees NOT to use tanning beds
7. Subject is willing to forego treatment of each Target cNF, except protocol specified therapy, during the study
8. Female subjects who are women of childbearing potential must have a negative urine pregnancy test result and be willing to use a protocol approved, contraceptive method for the duration of the study
9. Subject is willing and able to follow all study instructions and to attend all study visits.

Exclusion Criteria:

1. Subject has used any of the following topical therapies within the specified period prior to Visit 1 on or in proximity to any Target cNF that, in the investigator's opinion, impairs evaluation of any the cNFs or which exposes the subject to an unacceptable risk by study participation:

   * Corticosteroids; 30 days
   * Prescription retinoids (e.g., tazarotene, tretinoin, adapalene); 30 days
   * > 5% of an alpha-hydroxy acid (e.g., glycolic acid, lactic acid); 30 days
   * Fluorouracil; 30 days
   * Imiquimod; 30 days
   * LASER, light (e.g., intense pulsed light [IPL], photo-dynamic therapy [PDT]) or other energy-based therapy; 180 days
   * MEK inhibitor or BRAF inhibitor; ever.
2. The subject has used any of the following systemic medications therapies within the specified period prior to Visit 1:

   * Retinoids (e.g., etretinate, isotretinoin); 90 days
   * MEK inhibitors; 180 days
   * BRAF inhibitors; 180 days
3. Subject has a history of hypersensitivity to any of the ingredients in the study medications
4. Subject has any known intercurrent illness or physical condition that would, in the investigator's opinion, impair evaluation of a Target cNF or which exposes the subject to an unacceptable risk by study participation
5. Subject has, in the investigator's opinion, clinically relevant history of liver disease, including viral hepatitis, current alcohol abuse, or cirrhosis
6. Subject has a history of metastatic disease, or active cancer (excluding nonmelanoma skin cancer, Stage I cervical cancer, ductal carcinoma in situ of the breast, or Stage 0 chronic lymphocytic lymphoma) within the previous 5 years
7. Subject has any condition (e.g., other skin conditions or diseases, metabolic dysfunction, physical examination findings, clinical laboratory findings) or situation (e.g., vacation, scheduled surgery) that would, in the investigator's opinion, impair evaluation of a Target cNF or which exposes the subject to an unacceptable risk by study participation
8. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Safety and effectiveness of once daily NFX-179 gel treatment for 182 days measured by local tolerability assessments, safety laboratory tests, and target cNF volume reduction | 182 days
  Safety will be measured by routine safety laboratory tests (CBC/differential, serum chemistry, urinalysis), and local tolerability assessment where the investigator will assess erythema, edema, scabbing/crusting, vesiculation, and erosion. The subject will assess stinging, burning, and pruritus. All assessments are performed using a 4-point scale (0 none, 1 mild, 2 moderate, 3 severe). Effectiveness will be measured by the percent of treated subjects with at least a 50% reduction in cNF volume after 6 months of treatment.
Safety of once daily NFX-179 gel treatment for 182 days by adverse events and serious adverse events assessments | 182 days
  Safety of NFX-179 gel compared to the vehicle group will be measured by the assessment and occurrence of new and ongoing adverse events (AEs)/serious adverse events (SAEs).

SECONDARY OUTCOMES:
Percent of subjects with at least 50% Target cNF volume reduction after 182 days | 182 days
  Treatment effectiveness will be measured by the percent of treated subjects with at least a 50% reduction in cNF volume after 6 months of treatment. Tumor volume will be measured by ruler measurements and two-dimensional photography. All modes of tumor volume measurement are reported in cubic millimeters.
Percent change in cNF volume over 182 days | 182 days
  Percent change of tumor volume will be calculated through ruler measurements and two-dimensional photography throughout the course of treatment. All modes of tumor volume measurement are reported in cubic millimeters.
Physician's Tumor Assessment of Target cNF severity over 182 days | 182 days
  Effect of treatment with The Physician Tumor Assessment is the investigator's assessment of the average overall severity of each Target cNF tumor at a particular time point. The Physician Tumor Assessment is a 5-point measuring tumor severity (0 clear/none, 1 almost clear, 2 mild, 3 moderate, 4 severe). This assessment is performed at Screening, Baseline/Day 1, Days 58, 183, and 211.
Subject's Self-Assessment of Target cNF severity over 182 days | 182 days
  The Subject Self-Assessment is the subject's assessment of the average overall severity of each Target cNF at a particular time point and is not a comparison with any other time point. The Subject Self-Assessment is a 5-point measuring tumor severity (0 clear/none, 1 almost clear, 2 mild, 3 moderate, 4 severe). This assessment is performed at Screening, Baseline/Day 1, Days 58, 183, and 211.

OTHER OUTCOMES:
Patient Reported Outcome Measure to assess Target cNF symptoms over 182 days | 182 days
  This assessment is performed via the subject's assessment of their experience over the previous week with 9 items for each Target cNF (sensitivity, pain, itch, noticeability, size, appearance, care to avoid irritation, how much the cNF bothers the subject, self-consciousness). Each item is assessed by using a 5-point scale.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University Clinical Trials, Inc., San Diego, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Northshore University HealthSystem, Evanston, Illinois
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - The Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - Skin Specialists, P.C., Omaha, Nebraska
  - Sadick Research Group, LLC, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Apex Clinical Research Center, LLC, Mayfield Heights, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Derm Dox Center for Dermatology, Sugarloaf, Pennsylvania
  - Dermatology Treatment and Research Center, Dallas, Texas
  - UTHealth McGovern Medical School, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No